CLINICAL TRIAL: NCT03682068
Title: A Phase III, Randomized, Open-Label, Controlled, Multi-Center, Global Study of First-Line Durvalumab in Combination With Standard of Care Chemotherapy and Durvalumab in Combination With Tremelimumab and Standard of Care Chemotherapy Versus Standard of Care Chemotherapy Alone in Patients With Unresectable Locally Advanced or Metastatic Urothelial Cancer.
Brief Title: Study of Durvalumab Given With Chemotherapy, Durvalumab in Combination With Tremelimumab Given With Chemotherapy, or Chemotherapy in Patients With Unresectable Urothelial Cancer
Acronym: NILE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D933SC00001; 2018-001883-48 (EudraCT Number)
Record Dates: First submitted 2018-09-06; First posted 2018-09-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Locally Advanced Urothelial Cancer; Metastatic Urothelial Cancer
Keywords: renal pelvis; ureters; urinary bladder; urethra; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; tremelimumab; Cisplatin; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Durvalumab in Combination with SoC Chemotherapy (Experimental): Durvalumab every 3 weeks in concurrence with chemotherapy, followed by durvalumab monotherapy every 4 weeks.
  All patients will receive one of the following standard of care chemotherapy regimens every 3 weeks for 6 cycles:
  * cisplatin+ gemcitabine
  * If the patient is cisplatin-ineligible, carboplatin + gemcitabine
  Interventions: Drug: Durvalumab; Drug: Cisplatin + Gemcitabine; Drug: Carboplatin + Gemcitabine
- Durvalumab in Combination with Tremelimumab+SoC Chemotherapy (Experimental): Durvalumab and Tremelimumab every 3 weeks in concurrence with chemotherapy, followed by durvalumab monotherapy every 4 weeks
  Tremelimumab will be provided for 4 cycles.
  All patients will receive one of the following standard of care chemotherapy regimens every 3 weeks for 6 cycles:
  * cisplatin+ gemcitabine
  * If the patient is cisplatin-ineligible, carboplatin + gemcitabine
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Cisplatin + Gemcitabine; Drug: Carboplatin + Gemcitabine
- SoC Chemotherapy (Active Comparator): Patients will receive one of the following standard of care chemotherapy regimens every 3 weeks for 6 cycles:
  * cisplatin+ gemcitabine
  * If the patient is cisplatin-ineligible, carboplatin + gemcitabine
  Interventions: Drug: Cisplatin + Gemcitabine; Drug: Carboplatin + Gemcitabine

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion)
  Other Names: MEDI4736
  Arms: Durvalumab in Combination with SoC Chemotherapy; Durvalumab in Combination with Tremelimumab+SoC Chemotherapy
Drug: Tremelimumab — Tremelimumab IV (intravenous infusion)
  Arms: Durvalumab in Combination with Tremelimumab+SoC Chemotherapy
Drug: Cisplatin + Gemcitabine — Cisplatin IV (intravenous)+ Gemcitabine IV(intravenous), as standard of care.
Drug: Carboplatin + Gemcitabine — Carboplatin IV (intravenous)+ Gemcitabine IV(intravenous), as standard of care.

SUMMARY:
This is a randomized, open-label, controlled, multi-center, global Phase III study to determine the efficacy and safety of combining durvalumab ± tremelimumab with standard of care (SoC) chemotherapy (cisplatin + gemcitabine or carboplatin + gemcitabine doublet) followed by durvalumab monotherapy versus SoC alone as first-line chemotherapy in patients with histologically or cytologically documented, unresectable, locally advanced or metastatic transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary bladder, and urethra).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with histologically or cytologically documented, unresectable, locally advanced or metastatic transitional cell carcinoma (transitional cell and mixed transitional/non-transitional cell histologies) of the urothelium (including renal pelvis, ureters, urinary bladder, and urethra)
* Patients who have not been previously treated with first-line chemotherapy. Patients who have received prior definitive chemoradiation, adjuvant or neoadjuvant treatment for locally advanced disease are eligible provided that progression to locally advanced or metastatic disease has occurred >12 months from the last therapy [for chemoradiation and adjuvant treatment] or >12 months from the last surgery [for neoadjuvant treatment].
* At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion at baseline.
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at enrolment
* Adequate organ and marrow function as defined in the protocol
* Life expectancy ≥12 weeks in the opinion of the investigator
* Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients.

Key Exclusion Criteria:

* Prior exposure to immune-mediated therapy (with exclusion of Bacillus Calmette Guerin), including but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD L1, or anti-PD-L2 antibodies, except therapeutic anticancer vaccines, which are permitted. Prior local intervesical chemotherapy or immunotherapy is allowed if completed at least 28 days prior to the initiation of study treatment.
* No severe concomitant condition that requires immunosuppression medication
* Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* Patients who may be eligible for or are being considered for radical resection during the course of the study.
* Any medical contraindications to platinum (cisplatin or carboplatin) based doublet chemotherapy and/or known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | approximately 5 years
  OS is defined as the time from the date of randomization until death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) | approximately 5 years
  Additional analysis beyond the primary endpoint
Overall Survival at 24 months (OS24) | 24 months
  The OS24 will be defined as the Kaplan-Meier estimate of OS at 24 months
Progression Free Survival (PFS) | approximately 5 years
  PFS (per RECIST 1.1) will be defined as the time from the date of randomization until the date of first objective disease progression or death
Alive and Progression Free Survival at 12 months (APF12) | 12 months
  The APF12 will be defined as the Kaplan-Meier estimate of PFS (per RECIST 1.1) at 12 months
Objective Response Rate (ORR) | approximately 5 years
  ORR (per RECIST 1.1) is defined as the number (%) of patients with at least 1 visit response of complete response or partial response and will be based on a subset of all randomized patients
Duration of Response (DoR) | approximately 5 years
  DoR (per RECIST 1.1) will be defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression
Disease Control Rate (DCR) | approximately 5 years
  DCR is defined as the proportion of subjects with the best overall response of complete response, partial response or stable disease per RECIST 1.1
Time from randomization to second (PFS2) | approximately 5 years
  PFS2 will be defined as the time from the date of randomization to the earliest of the progression events subsequent to that used for the PFS endpoint or death
To assess disease-related symptoms, physical functioning, and other Health-related quality of life | approximately 5 years
  Collection of patient reported outcome questionnaires

OTHER OUTCOMES:
To assess safety using a summary of adverse events. | approximately 5 years
  Adverse Events (both in terms of MedDRA preferred terms and CTCAE grade) will be listed individually by patient. The number of patients experiencing each Adverse Event will be summarized by treatment arm and CTCAE grade
To assess pharmacokinetics of Durvalumab and Tremelimumab | approximately 5 years
  Serum concentrations of Durvalumab and Tremelimumab
To assess immunogenicity of Durvalumab and Tremelimumab | approximately 5 years
  Presence of anti-drug antibodies for Durvalumab and Tremelimumab

CONTACTS AND LOCATIONS:
Locations (173):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Salinas, California
  - Research Site, Santa Barbara, California
  - Research Site, Truckee, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Orlando, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Grand Rapids, Michigan
  - Research Site, Bozeman, Montana
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Germantown, Tennessee
  - Research Site, Fort Worth, Texas
- Argentina (2):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
- Australia (8):
  - Research Site, Box Hill
  - Research Site, Elizabeth Vale
  - Research Site, Kogarah
  - Research Site, Macquarie University
  - Research Site, Murdoch
  - Research Site, Orange
  - Research Site, South Brisbane
  - Research Site, St Albans
- Brazil (9):
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (17):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Szolnok
- India (8):
  - Research Site, Gūrgaon
  - Research Site, Hubli
  - Research Site, Kolkata
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Pune
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (9):
  - Research Site, Arezzo
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Terni
  - Research Site, Verona
- Japan (20):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Kanazawa
  - Research Site, Kita-gun
  - Research Site, Koshigaya-shi
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Miyazaki
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Toyama
  - Research Site, Yokohama
- Philippines (7):
  - Research Site, Bacolod
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Radom
  - Research Site, Warsaw
- Russia (9):
  - Research Site, Ivanovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Omsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Tyumen
  - Research Site, Vologda
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santander
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Mueang
  - Research Site, Songkhla
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home